CLINICAL TRIAL: NCT05726422
Title: Use of a 10 Points Visual Analogue Food Intake Scale for Children to Assess Intake: Prospective Study
Acronym: CESAR
Status: Terminated | Type: Observational
Why Stopped: Sufficient number of subjects included for analyzes
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0308; 2022-A01448-35 (Other: ANSM)
Record Dates: First submitted 2023-01-19; First posted 2023-02-14 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-08

CONDITIONS: Child Malnutrition
Keywords: children; undernutriton; food intake
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In hospitalized children, undernutrition increases the length of hospitalization, aggravates the causal pathology, favors the occurrence of complications, and increases the cost of hospitalization. With a prevalence of 10 to 20%, undernutrition is therefore a major problem which, moreover, is largely under-diagnosed.

The evaluation of food intake has historically been based on the evaluation of food consumption by means of a food card or a food survey during the last 24 hours.

In adults, a rapid assessment tool has been developed, the SEFI® (Score Evaluation Facile des Ingestats), consisting of a visual analog scale (VAS) graduated from 0 to 10. It has been validated as being concordant with previous tools for the assessment of dietary intake in the general population and is now recommended for adults. It allows early identification of a risk of undernutrition when the score is < 7/10.

We propose to evaluate the correlation between this 10-point analog scale (SEFI) and ingesta in children in relation to recommended energy intakes for age and weight.

DETAILED DESCRIPTION:
Data collection at the foot of the bed during hospitalization or after the consultation on a data collection form.

Conventional admission of patients to the departments involved. Carrying out the study (questionnaire and measurements) in the room. It will not be necessary to move the patients. The weighing and measuring of patients is not different from the usual care carried out during an admission to hospital in the services concerned by the study. All anthropometric measurements correspond to the recommendations of good practice. Anthropometric measurements will be performed by the health care team.

The dietary survey will be carried out by a dietician from the UTN or the pediatric team with an evaluation of the caloric intake at the time. The results will then be entered into the GENI software using the CIQUAL table in order to calculate the caloric intake (and the composition of trace elements and vitamins) according to standardized tables of food composition. The child will be accompanied by his or her parents for this survey.

The child will be asked the following question: "On a scale of 0 to 10, if 0 is "in terms of quantity, I don't eat anything at all" and 10 is "I eat as usual", between 0 and 10 where do you stand today? The same question will be asked of the parent. The parent will be blind to the child's response.

Blinding between the different assessments will be maintained as follows: the dietary survey will be conducted by a dietician blind to the SEFI scores, and the SEFI will be administered to the child and parents separately, by 2 different blind operators (childcare workers or assistant childcare workers), themselves blind to the dietary survey.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 6 months to less than 18 years
* Patient admitted in short and long stay pediatric services at the Montpellier University Hospital, other than maternity, neonatality, palliative care or intensive care, excluding SSR.
* Patient admitted for day hospitalization or consultation at the Montpellier University Hospital

Exclusion Criteria:

* Opposition from parents or child
* Pathology involving the satiety centers
* Breast-fed child
* Proven disorder of orality
* Strict fasting by the medical team
* Anorexia nervosa
* Consciousness disorder
* Exclusive artificial feeding

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children admitted for hospitalization or consultation during the study period until the required number of subjects was obtained.
  300 subjects 150/150 : hospitalisation/consultation
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
To assess the diagnostic validity of the SEFI, a 10-item self-administered numerical scale assessing food intake, for the diagnosis of decreased ingesta in children. | At the inclusion
  Concordance between a Probationary Test and a Reference Test:
  Probationary test
  Verbal assessment of ingesta by the SEFI, administered orally to the patient. the thresholds that will be tested is <7/10.
  Reference test Ingesta representing at least 2/3 of recommended ingesta. Ingesta is assessed by a 24-hour recall performed by a dietician with children, accompanied by their parents.
To assess the diagnostic validity of the SEFI, a 10-item self-administered numerical scale assessing food intake, for the diagnosis of decreased ingesta in children. | At the inclusion
  Concordance between a Probationary Test and a Reference Test:
  Probationary test
  Verbal assessment of ingesta by the SEFI, administered orally to the patient. the thresholds that will be tested is <10/10.
  Reference test Ingesta representing at least 2/3 of recommended ingesta. Ingesta is assessed by a 24-hour recall performed by a dietician with children, accompanied by their parents.

SECONDARY OUTCOMES:
Measure of percentage of ingesta against recommended ingesta | At the inclusion
  Concordance between a Probationary Test and a Reference Test:
  Probationary test
  Verbal assessment of ingesta by the SEFI, administered orally to the patient.
  Reference test: the percentage of caloric consumption in relation to the recommended ingesta according to age.
Measure of undernutrition in children with the SEFI <7/10 | At 4 months (end of the recruitment period)
  Concordance between a Probationary Test and a Reference Test:
  Probationary test
  Verbal assessment of ingesta by the SEFI, administered orally to the patient. The thresholds that will be tested is <7/10.
  Reference test: Diagnosis of undernutrition according to the HAS 2019.
Measure of nutritional deficiencies in the diet | At the inclusion
  Concordance between a Probationary Test and a Reference Test:
  Probationary test
  Verbal assessment of ingesta by the SEFI, administered orally to the patient.
  Reference test: Nutrition deficeinies in the diet according to international recommendations for children's intakes
Concordance of the SEFI administered to children and the SEFI administered to parents | At the inclusion
  Concordance between a Probationary Test and a Reference Test:
  Probationary test
  Verbal assessment of ingesta by the SEFI, administered orally to the patient.
  Reference test: Verbal assessment of ingesta by the SEFI, administered orally to the parents.
Number of children's responses to the SEFI according to age | At the inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier - Hôpital Lapeyronie, Montpellier, France

REFERENCES:
- [Background] Hankard R, Colomb V, Piloquet H, Bocquet A, Bresson JL, Briend A, Chouraqui JP, Darmaun D, Dupont C, Frelut ML, Girardet JP, Goulet O, Rieu D, Simeoni U, Turck D, Vidailhet M. [Malnutrition screening in clinical practice]. Arch Pediatr. 2012 Oct;19(10):1110-7. doi: 10.1016/j.arcped.2012.07.024. Epub 2012 Sep 5. French. PMID 22959889
- [Background] Diagnostic de la dénutrition de l'enfant et de l'adulte [Internet]. Haute Autorité de Santé. [cited 2021 May 24]. Available from: https://www.has-sante.fr/jcms/p_3118872/fr/diagnostic-de-la-denutrition-de-l-enfant-et-de-l-adulte
- [Background] Thibault R, Goujon N, Le Gallic E, Clairand R, Sebille V, Vibert J, Schneider SM, Darmaun D. Use of 10-point analogue scales to estimate dietary intake: a prospective study in patients nutritionally at-risk. Clin Nutr. 2009 Apr;28(2):134-40. doi: 10.1016/j.clnu.2009.01.003. Epub 2009 Feb 14. PMID 19223093
- [Background] Guerdoux-Ninot E, Flori N, Janiszewski C, Vaille A, de Forges H, Raynard B, Baracos VE, Thezenas S, Senesse P. Assessing dietary intake in accordance with guidelines: Useful correlations with an ingesta-Verbal/Visual Analogue Scale in medical oncology patients. Clin Nutr. 2019 Aug;38(4):1927-1935. doi: 10.1016/j.clnu.2018.06.974. Epub 2018 Jun 30. PMID 30355527
- [Background] De Longueville C, Robert M, Debande M, Podlubnai S, Defourny S, Namane SA, Pace A, Brans C, Cayrol E, Goyens P, De Laet C. Evaluation of nutritional care of hospitalized children in a tertiary pediatric hospital. Clin Nutr ESPEN. 2018 Jun;25:157-162. doi: 10.1016/j.clnesp.2018.02.008. Epub 2018 Mar 14. PMID 29779812